CLINICAL TRIAL: NCT05885945
Title: Diaphragmmatic Muscle Strength and Balance in Women With Dysmenorhea
Acronym: Dysmenorhea
Status: Completed | Type: Observational
Sponsor: Catholic University of Murcia (Other)
Responsible Party: Principal Investigator, Felipe León Morillas, Dr., Catholic University of Murcia
Other Study IDs: TC-01/23
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Dysmenorrhea Primary
Keywords: dysmenorrhea; diaphragm; balance; muscular strength
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dysmenorrhea: primary dysmenorrhea
- control: control not pain

SUMMARY:
Analysis of stabilometric and respiratory variables in patients with dysmenorrhea during the first day of the menstrual cycle and any other day outside the cycle.

DETAILED DESCRIPTION:
Sociodemographic variables such as age, height, body mass index.

Respiratory variables such as maximum inspiratory pressure (MIP), MIP reference %, and MIP predictive value.

Stabilometric variables we will measure the balance in condition of eyes open and eyes closed bipodal support and eyes open in monopodal support

ELIGIBILITY:
Inclusion Criteria:

* Adult women with primary dysmenorrhea.
* Not having had any type of childbirth (natural, caesarean section, etc).
* Not be positive in COVID. Antigen test in the last 24 hours or negative PCR in the last 48 hours.

Exclusion Criteria:

* Receive medical treatment during research.
* Have any orthopedic, neurological or systemic disease diagnosed other than primary dysmenorrhea.
* Be in follow-up with any medical treatment that does not be primary dysmenorrhea
* Women with a history of trauma or surgical treatment who involve the musculoskeletal system in the last year.
* Use of analgesics in the last 48 hours.
* Consumption of alcohol in the last 24 hours.
* Have a history or suspicion of pregnancy.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — WOMEN WITH PERIOD PAIN
Study Population: Women with primary dysmenorrhea
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Balance | 2 months
  stabilometric variables in bipodal and monopodal support
diaphragmatic muscle strength | 2 months
  diaphragmatic muscle force through the maximum inspiratory pressure in the mouth

SECONDARY OUTCOMES:
sociodemographic variables | 2 monsths
  sociodemographic variables such as age, body mass index, personal data record, and data record related to pain and dysmenorrhea

CONTACTS AND LOCATIONS:
Overall Officials: Felipe León-Morillas, Principal Investigator — Catholic University of Murcia
Locations (1):
- University Catholic of Murcia, Guadalupe, Murcia, Spain